CLINICAL TRIAL: NCT07392983
Title: Comparison of Effect of Dexmedetomidine and Midazolam on Emergence Agitation in Patients Undergoing Functional Endoscopic Sinus Surgery
Brief Title: Comparison of Effect of Dexmedetomidine and Midazolam on Emergence Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Madiha-BVH
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-D (Experimental): Patients were given a dexmedetomidine injection with a loading dose of 1 µg/kg in 10 minutes prior to the procedure.
  Interventions: Drug: Dexmedetomidine
- Group-M (Experimental): Patients received a midazolam injection with a loading dose of 0.02 mg/kg in 10 min prior the procedure.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Patients were given dexmedetomidine injection with a loading dose of 1 µg/kg in 10 minute prior to the procedure.
  Arms: Group-D
Drug: Midazolam — Patients received midazolam with a loading dose of 0.02 mg/kg in 10 min prior to the procedure.
  Arms: Group-M

SUMMARY:
Since the frequency of emergence agitation (EA) is relatively high in children while undergoing nasal surgery, and there is not much data available in Pakistan regarding EA in adults undergoing functional endoscopic sinus surgery (FESS). Hence there is a need to conduct this study in the local population to see the effect of dexmedetomidine and midazolam on EA. Therefore, the current study was initiated, aiming to compare the effect of dexmedetomidine and midazolam on EA in patients undergoing FESS.

DETAILED DESCRIPTION:
There is not much local data present on the topic of EA. As the frequency of EA is relatively high, it can lead to any unwanted event, which can lead to other complications in the patients undergoing nasal surgery. Although in some studies dexmedetomidine has been found to significantly reduce the frequency of EA and severity, provide better sedation, and lower the need for postoperative rescue analgesia in patients undergoing FESS, few others have claimed comparable results for midazolam as well. The findings of this study would not only add to the local data but also be helpful in determining a better option in reducing the frequency of this phenomenon in patients undergoing FESS under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 16-60 years
* Undergoing elective FESS under general anesthesia

Exclusion Criteria:

* Patients with the presence of infection at the site of the blockage
* Epilepsy, myasthenia gravis, or polio (as per history and clinical record)
* Systemic illness (such as cardiac, hepatic, endocrinal or neurological)
* Substance induced disorder
* Psychiatric disorders
* Taking medications, such as alpha 2 agonists, beta blockers' or tricyclic anti-depressants
* Allergies to the medications used

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness in emergence agitation | 90 minutes
  The effectiveness of the treatment was assessed through Ricker's sedation and agitation score, with a score of 4 as efficacy 'yes'.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ashraf, Principal Investigator — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur; Ambreen Khan, FCPS, Study Director — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur
Locations (2):
- Pakistan (2):
  - Bahawal Victoria Hospital/Quad-e-Azam Medical College, Bahawalpur, Punjab Province
  - Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.